CLINICAL TRIAL: NCT00763295
Title: Is Tuberculin Skin Testing Effective in Screening for Latent Tuberculosis in Patients With HIV?
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Jordan Glaser, MD, Staten Island University Hospital
Other Study IDs: 08-015
Record Dates: First submitted 2008-09-28; First posted 2008-09-30 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Latent Tuberculosis; HIV Infections
Keywords: latent tuberculosis; HIV; IFN-γ based assay
MeSH Terms: conditions — Latent Tuberculosis; HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV infection
  Interventions: Other: T-Spot.TB test

INTERVENTIONS:
Other: T-Spot.TB test — diagnostic test

SUMMARY:
HIV infection highly increases the risk of progression of latent tuberculosis (TB) to active disease that therapy is recommended for all PPD-positive, HIV-infected patients, regardless of age. Sensitivity of the PPD testing is, however, dependent on a normal T cell function.

Therefore, an accurate and reliable method for detection of latent tuberculosis in patients with HIV is urgently needed.

This prospective study will examine the utility of interferon-gamma (IFN-γ) based assay, T-SPOT.TB,for detection of TB in HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria

* adult individuals with confirmed HIV infection

Exclusion Criteria:

* Patients who are on INH treatment
* Patients who have a positive PPD test within 1 year of study enrollment
* Individuals with blistering or ulcerating skin disorder
* Pregnant women
* Patients who were given blood transfusion within 6 weeks prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with HIV confirmed by standard methods
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States